CLINICAL TRIAL: NCT06123104
Title: Assessment of Automatic Tourniquets for Soldiers During Wartime as Part of Accelerated Research and Development
Brief Title: Assessment of Automatic Tourniquets for Soldiers During Wartime
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical Corps, Israel Defense Force (Other)
Responsible Party: Principal Investigator, TOMER ERLICH, Head of Innovation, R&D Directorate, IDF Medical Corps Head of Medical Research, Directorate of Defense R&D, Israeli Ministry of Defense (IMOD DDR&D), Medical Corps, Israel Defense Force
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 1.1
Record Dates: First submitted 2023-10-31; First posted 2023-11-08 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Trauma Injury; Hemorrhage Wound
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Automatic Tourniquet (Experimental): Automatic pneumatic tourniquet
  Interventions: Device: Occlusion of blood flow diagnosed by Point of Care UltraSound (POCUS)
- Combat Application Tourniquet (CAT) (Active Comparator): Combat Application Tourniquet Generation 7
  Interventions: Device: Occlusion of blood flow diagnosed by Point of Care UltraSound (POCUS)

INTERVENTIONS:
Device: Occlusion of blood flow diagnosed by Point of Care UltraSound (POCUS) — Tourniquets will be applied until peripheral blood flow occlusion is achieved. Total intervention time: up to 60 seconds

SUMMARY:
The goal of this clinical trial is to compare usability and performance of automatic tourniquets (AUT) and standard mechanical tourniquets (CAT) in healthy adults. The main questions it aims to answer are:

* Are AUTs effective in occlusion of blood flow
* Are AUTs easy to use

Participants will be asked to place AUT and CAT on their upper limbs and lower limbs (8 applications overall).

Following each application, the following parameters will be assessed:

1. Limb blood flow
2. Ease of use

Researchers will compare the results of the AUT and CAT to see if AUT is as effective as CAT in blood occlusion, and if AUT is easy to use as the CAT.

DETAILED DESCRIPTION:
The goal of this clinical trial is to compare usability and performance of automatic tourniquets (AUT) and standard mechanical tourniquets (CAT) in healthy adults. The main questions it aims to answer are:

* Are AUTs effective in occlusion of blood flow
* Are AUTs easy to use

Participants will be asked to place AUT and CAT on their upper limbs and lower limbs (8 applications overall).

ELIGIBILITY:
Inclusion Criteria:

-Soldier in active service or active reserve service.

Exclusion Criteria:

* Muscle disorders
* Peripheral nerve disorders
* Skin diseases of the limbs
* Limb surgery in the past
* Rickets
* Hypertension

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-10-27 (Actual); Primary Completion 2024-11-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to distal limb arterial occlusion as assessed by Doppler | 60 seconds
  Time to distal limb arterial occlusion as assessed by Doppler is recorded

SECONDARY OUTCOMES:
Safety of using automatic tourniquets | Will be assessed via questionnaire up to 5 minutes following the intervention.
  Safety issues, specifically peripheral limb numbness will be assessed via questionnaire. Scale is from 0 to 5, 0 is "No numbness", 5 is "Severe numbness"
Usability of using automatic tourniquets | Ease of use will be assessed via questionnaire up to 5 minutes following the intervention.
  Usability of using automatic tourniquets will be assessed via questionnaire up to 5 minutes following the intervention. Scale for ease to secure the tourniquet is from 0 to 5, 0 is "Very difficult to secure", 5 is "Very easy to secure"

CONTACTS AND LOCATIONS:
Overall Officials: Tomer Erlich, MD, Principal Investigator — Head of Medical innovation and R&D
Locations (1):
- Tel hashomer, Ramat Gan, Israel